CLINICAL TRIAL: NCT02134379
Title: Dynamic Thoracic Impedance as a Marker for Heart Failure Decompensation: A Pilot Trial of the "Dynamic Thoracic Impedance Bed Rest Test"
Brief Title: Dynamic Thoracic Impedance as a Marker for Heart Failure Decompensation
Status: Completed | Type: Observational
Sponsor: Charles Porter, MD (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Charles Porter, MD, Clinical Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: STUDY00000596
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure; With Decompensation
Keywords: Thoracic Impedance; Diagnostic Marker; Bed Rest Test; Transthoracic Impedance; Heart Failure; HF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: Subjects have implanted Medtronic device and a primary diagnosis of left ventricular systolic dysfunction
  Interventions: Device: Medtronic ICDs, CRT-Ds, and CRT-Ps

INTERVENTIONS:
Device: Medtronic ICDs, CRT-Ds, and CRT-Ps — Any Medtronic implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT) device. Device must have capacity to measure thoracic impedance as described in protocol. This includes the majority of FDA-approved Medtronic devices currently in use.
  Other Names: ICDs:; Evera(TM) XT DR (Models DDBB1D4, DDBB1D1); Evera(TM) XT VR (Models DVBB1D4, DVBB1D1); Protecta(R) XT DR (Models D314DRG, D314DRM); Protecta(R) XT VR (Models D314VRG, D314VRM); Secura(R) DR (Models D224DRG, D204DRM); Secura(R) VR (Models D224VRC, D204VRM); Virtuoso(R) II DR (Model D274DRG); Virtuoso(R) II VR (Model D274VRC); Virtuoso(R) DR (Model D154AWG); Virtuoso(R) VR (Model D154VWC); CRT-Ds/CRT-Ps:; Viva(TM) XT CRT-D (Models DTBA1D1, DTBA1D4); Viva(TM) S CRT-D (Models DTBB1D1, DTBB1D4); InSync Sentry(R) CRT-D (Models 7297, 7299); Protecta(R) XT CRT-D (Models D314TRM, D314TRG); Concerto(R) II CRT-D (Model D274TRK); Consulta(R) CRT-D (Models D204TRM, D224TRK); Concerto(R) CRT-D (Models C154DWK, C164AWK); Consulta(R) CRT-P (Model C4TR01)

SUMMARY:
This pilot study proposes to perform measurements of approved thoracic impedance technology that will help answer questions in patients with decompensated heart failure.

DETAILED DESCRIPTION:
Improved metrics derived from the transthoracic impedance (Z) available from implanted Medtronic devices may provide more sensitive indicators of the state of compensation for heart failure patients. Quantification of specific data may provide new information that can improve quality of life for patients and offer vital information to clinicians regarding the adequacy of inpatient and outpatient assessment and management of acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systolic dysfunction
* Able to provide informed consent
* Have a Medtronic manufactured device with Thoracic Impendence Monitoring capabilities

Exclusion Criteria:

* Patients with severe congestive heart failure who are intubated
* Patients who are oxygen dependent on continuous positive or bilevel positive ventilation
* Inability to tolerate postural variations due to congestive heart failure or other medical or surgical condition.Unable to complete proposed testing
* Subjects who cannot giveWill not give written, informed consent on their own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified from the KU Hospital Cardiology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from sitting to supine to standing in thoracic impedance | Baseline, 30 Days
  thoracic impedance will be measured at each position at baseline visit then again at the follow-up visits through 30 days

SECONDARY OUTCOMES:
Rate of change in thoracic impedance | Baseline, 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Porter, MD, FACC, FACP, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States